CLINICAL TRIAL: NCT06619743
Title: Study on HPV Infection and Vaginal Microecology in Immunosuppressed Women
Brief Title: HPV Infection and Vaginal Microecology in Immunosuppressed Women
Status: Not yet recruiting | Type: Observational
Sponsor: Lan Zhu (Other)
Responsible Party: Sponsor-Investigator, Lan Zhu, Director of the Department of Obstetrics and Gynecology at Peking Union Medical College Hospital, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Other Study IDs: K6758
Record Dates: First submitted 2024-09-27; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: HIV Infections; HPV Infection; Cervical Cancer; Anal Cancer
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections; Uterine Cervical Neoplasms; Anus Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to establish a screening cohort for HPV infection and related tumors in areas with high incidence of HIV infection, explore the screening of cervical cancer and anal cancer and the prognosis management model of precancerous lesions in HIV-infected women, and provide a scientific basis for the formulation of malignant tumor screening policies for this population in my country. In addition, this study intends to characterize the cervical, vaginal, and intestinal microecological characteristics of women with different HIV/HPV infection status, so as to explore the impact of cervical, vaginal, and intestinal microecological characteristics on persistent HPV infection or CIN/cancer progression.

ELIGIBILITY:
Inclusion Criteria:

* HIV positive female, ≥18 years old
* HIV infection is sexually transmitted
* Have an intact cervix
* Have not received cervical cancer screening in the past 1 year
* No previous treatment for CIN/cervical cancer
* No clinical pregnancy symptoms

Exclusion Criteria:

* Women who have had a previous cervical resection
* Unable to complete all screening processes independently
* Unable or unwilling to accept follow-up
* For subjects in vaginal microecology studies, women who used antibiotics within 2 weeks before collecting vaginal secretions, had sexual intercourse within 3 days, or used vaginal medication or vaginal douching within 48 hours need to be further excluded.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected women
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection rate of cervical intraepithelial neoplasia grade 2 or above (CIN2+) in women infected with HIV within 5 years | 5 years
  Detection rate of cervical intraepithelial neoplasia grade 2 or above (CIN2+) in women infected with HIV within 5 years
Detection rate of cervical intraepithelial neoplasia grade 3 and above (CIN3+) in women infected with HIV within 5 years | 5 years
  Detection rate of cervical intraepithelial neoplasia grade 3 and above (CIN3+) in women infected with HIV within 5 years

IPD SHARING:
Plan to Share IPD: No